CLINICAL TRIAL: NCT04653532
Title: Mobile Health Biometrics to Enhance Exercise and Physical Activity Adherence in Type 2 Diabetes: A Pilot Randomized Trial
Brief Title: Mobile Health to Enhance Exercise in Type 2 Diabetes
Acronym: MOTIVATET2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Liverpool John Moores University (Other); University of Exeter (Other); Medical Research Council (Other Government); Lancaster University (Other)
Responsible Party: Principal Investigator, Jonathan Little, associate professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20-01936; 20/SS/0101 (Other: South East Scotland Research Ethics Committee)
Record Dates: First submitted 2020-11-19; First posted 2020-12-04 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 2; Telemedicine; Mobile Applications; Exercise Therapy
Keywords: Humans; Blood Glucose; Exercise; Life Style; Counseling; Biomedical Technology
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth Technology (Experimental): Participants in this group (Mobile health technology (mHealth)) will receive the same 6-month exercise and physical activity programme supported by an exercise specialist, but participants in this group will also receive a fitness watch that links to a mobile phone application (App).
  Interventions: Behavioral: Exercise Programme and Counselling; Device: Polar Ignite and App
- Exercise Counselling (Active Comparator): Participants in this group (Exercise Counselling) will complete a 6-month structured exercise and physical activity programme supported by regular contact with an exercise specialist.
  Interventions: Behavioral: Exercise Programme and Counselling

INTERVENTIONS:
Behavioral: Exercise Programme and Counselling — A 6 month exercise and physical activity programme supported by an exercise specialist
Device: Polar Ignite and App — A fitness watch that links to a mobile phone application (App) which enables the exercise specialist to provide greater support and feedback throughout the programme
  Other Names: Polar Watch; Polar Flow
  Arms: mHealth Technology

SUMMARY:
Being physically active and exercising is important for the treatment of Type 2 diabetes as it helps control blood sugar and improve physical function. Lots of people find it hard to be physically active and sticking with exercise is difficult for most people. In this project we will investigate two strategies to support people with Type 2 diabetes to increase and then maintain a physically active lifestyle, which includes exercising regularly. Participants in one group (Exercise Counselling) will complete a 6-month structured exercise and physical activity programme supported by regular (virtual) contact with an exercise specialist. Participants in the second group (Mobile health technology (mHealth)) will receive the same 6-month exercise and physical activity programme supported by an exercise specialist, but participants in this group will also receive a fitness watch that links to a mobile phone application (App). The fitness watch and mobile App will allow the exercise specialist to provide greater support and feedback throughout the programme.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2D within the previous 5-24 months
* Male or Female
* Aged 40-75
* Treat diabetes with only Metformin or lifestyle modifications (diet and exercise)
* For those prescribed Metformin: have used a stable dose for 3-months or more

Exclusion Criteria:

* Aged under 40 or over 75
* Glycated hemoglobin level (HbA1c) more than 10% (>86mmol/mol)
* Blood pressure higher than 160/110 mmHg
* Treat diabetes with an antidiabetic drug other than Metformin (Sulfonylureas, Thiazolidinedione, dipeptidylpeptidase-4 inhibitors, sodium glucose co-transporter 2 inhibitors, glucagon-like peptide-1 receptor agonist, Acarbose, meglitinides)
* Prescription of Insulin
* Unstable angina (frequent chest pain)
* Myocardial infarction (heart attack) within the previous 3 months
* Transient ischemic attack (TIA) within the previous 6 months
* Heart failure ≥class 2
* Arrhythmia
* Inability to increase activity
* Pregnancy or planning to become pregnant
* Less than 6 months post childbirth or stopped breastfeeding less than 1 month ago
* Not owning a smartphone/ or having no data plan or access to WiFi
* currently meeting the recommended exercise guidelines (150 min of moderate intensity exercise per week).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Determine the number of adults with newly diagnosed T2D that are eligible to participate in the trial | 0-12 months
  Information will be collected on:
  - The number of patients approached and reasons for not joining the study
The number of these adults with newly diagnosed T2D who would be willing to take part in this trial | 0-12 months
  Information will be collected on:
  - The number of patients who actually enroll
The characteristics of these adults with newly diagnosed T2D who are willing to take part in the trial | 0-12 months
  Information will be collected on:
  - Patient gender, age, and how patients are currently treating their T2D
The number and percentage of participants retained at 12-months. | 0-12 months
  Information will be collected on:
  - Number and percentage of patients attending at 12-month follow up and reasons for drop-out.

SECONDARY OUTCOMES:
Adherence to exercise | 0 months, 0-6 months, 0-12 months
  Adherence to structured exercise assessed through monthly exercise questionnaire (GLTEQ)
Change in glycaemic control | 0 months, 0-6 months, 0-12 months
  Glycated hemoglobin (HbA1c), flash glucose monitoring
Change in body composition | 0 months, 0-6 months, 0-12 months
  Height (meters) and weight (kilograms) will be aggregated to arrive at one reported BMI value (kg/m^2)
Change in weight | 0 months, 0-6 months, 0-12 months
  Weight (kilograms)
Change in waist circumference | 0 months, 0-6 months, 0-12 months
  Waist circumference (centimeters)
Change in blood pressure | 0 months, 0-6 months, 0-12 months
  Blood pressure taken with a cuff
Change in blood lipids | 0 months, 0-6 months, 0-12 months
  Total cholesterol, high-density lipoprotein, triglycerides, low-density lipoprotein
Diabetes related quality of life | 0 months, 0-6 months, 0-12 months
  SF-12 Health Survey and Diabetes Treatment Satisfaction Questionnaire used to assess diabetes related quality of life
Behavioural regulation in exercise | 0 months, 0-6 months, 0-12 months
  Assessed using the Behavioural Regulation in Exercise Questionnaire
Patient rapport with counsellor | 0 months, 0-6 months, 0-12 months
  Assessed using the Patient Rapport with Counsellor Questionnaire

OTHER OUTCOMES:
Acceptability and feasibility of the wearable intervention to patients | 0-6 months, 0-12 months
  Post-intervention patient questionnaire that will assess the acceptability of the wearable intervention and exposure to other wearable technologies
Acceptability and feasibility of patients continuing the intervention on their own | 0-6 months, 0-12 months
  Follow-up patient questionnaire investigating anticipated barriers and facilitators to continuing the intervention
Pilot methods for collecting outcome measures | Approx. 1 month after baseline
  Early acceptability questionnaire investigating the acceptability of the measurement instruments and their ease of use.
Ensure that our plans for recruitment, randomisation, treatment, and follow-up are acceptable to patients | 0-12 months
  Post intervention patient questionnaire investigating the acceptability of the recruitment and randomisation process and the measurement instruments
Determine availability and completeness of economic data | 0 months, 0-6 months, 0-12 months
  5-level EQ-5D Questionnaire
Determine healthcare usage | 0 months, 0-6 months, 0-12 months
  Questionnaire assessing healthcare usage in the last 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymised data from this study will be made available for sharing with other investigators, after publication of the study's key papers. Data will be shared through the LJMU Data Repository (http://opendata.ljmu.ac.uk/). This is a secure institutional data repository, which is searchable on the www, it is managed by Library Services. A DOI will be generated for datasets as they are deposited to the repository. Data will be stored in this repository for a minimum of 10 years or for 10 years from the last date of access.
Time Frame: Data will be stored in this repository for a minimum of 10 years or for 10 years from the last date of access.
Access Criteria: Data will be shared through the LJMU Data Repository (http://opendata.ljmu.ac.uk/). This is a secure institutional data repository, which is searchable on the www, it is managed by Library Services. A DOI will be generated for datasets as they are deposited to the repository.
URL: http://opendata.ljmu.ac.uk/

REFERENCES:
- [Derived] Low JL, Hesketh K, Falkenhain K, Jung ME, Singer J, Jones CA, Russon C, Cocks M, McManus A, Little JP; MOTIVATE T2D Team. Improved Glycemic Control in Adults with Type 2 Diabetes is More Strongly Associated with Exercise Duration Than with Volume, Frequency, or Consistency. Med Sci Sports Exerc. 2025 Dec 16. doi: 10.1249/MSS.0000000000003922. Online ahead of print. PMID 41398622
- [Derived] Hesketh K, Low J, Andrews R, Jones CA, Jones H, Jung ME, Little J, Mateus C, Pulsford R, Singer J, Sprung VS, McManus AM, Cocks M. Mobile Health Biometrics to Enhance Exercise and Physical Activity Adherence in Type 2 Diabetes (MOTIVATE-T2D): protocol for a feasibility randomised controlled trial. BMJ Open. 2021 Nov 26;11(11):e052563. doi: 10.1136/bmjopen-2021-052563. PMID 34836904